CLINICAL TRIAL: NCT02636699
Title: A Double-blind, Placebo-controlled, Randomized Phase 3 Pivotal Trial to Assess the Efficacy and Safety of Peanut Epicutaneous Immunotherapy With Viaskin Peanut in Peanut-allergic Children
Brief Title: Efficacy and Safety of Viaskin Peanut in Children With Immunoglobulin E (IgE)-Mediated Peanut Allergy
Acronym: PEPITES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEPITES
Record Dates: First submitted 2015-11-19; First posted 2015-12-22 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viaskin Peanut 250mcg (Experimental): One Viaskin epicutaneous delivery system (patch) containing 250 µg of peanut protein applied on the skin for 24 hours (±4 hours of allowance) daily for a period of 12 months.
  Interventions: Biological: Viaskin Peanut 250mcg
- Placebo (Placebo Comparator): One Viaskin epicutaneous delivery system (patch) containing placebo applied on the skin for 24 hours (±4 hours of allowance) daily for a period of 12 months.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Viaskin Peanut 250mcg — Peanut extract cutaneous patch
  Other Names: DBV712
  Arms: Viaskin Peanut 250mcg
Biological: Placebo — Cutaneous patch containing an inactive deposit manufactured to mimic peanut extract
  Arms: Placebo

SUMMARY:
The PEPITES study evaluates the efficacy and safety of Viaskin Peanut 250 µg peanut protein to induce desensitization to peanut in peanut-allergic children 4 through 11 years of age after a 12-month treatment by epicutaneous immunotherapy (EPIT).

DETAILED DESCRIPTION:
This is a 12-month, Phase III, double-blind, placebo-controlled, randomized study to assess the efficacy and safety of Viaskin Peanut, dosed at 250µg peanut protein (per patch) in peanut-allergic children from 4 through 11 years of age.

The overall maximum study duration for each subject is approximately 61 weeks (6-week screening period, 12-month treatment period and 2-week follow-up period).

During the screening period, subjects will undergo a first screening visit and an entry double-blind, placebo-controlled food challenge (DBPCFC) to peanut to confirm their allergy and their entry peanut eliciting dose (ED). The starting dose of the challenge will be 1 mg peanut protein and will escalate up to a highest dose of 300mg peanut protein. Subjects who react at or below the dose of 300mg peanut protein are considered eligible.

Randomization of eligible subjects will occur in a 2:1 ratio to Viaskin Peanut dosed at 250µg peanut protein (active treatment) or placebo. Subjects will be stratified at randomization by their entry/screening DBPCFC ED in 1 of the following 2 strata and by study center:

* Stratum 1: children with a screening ED of 1mg, 3mg or 10mg;
* Stratum 2: children with a screening ED of 30mg, 100mg or 300mg.

Subjects will apply a Viaskin patch containing either peanut protein or placebo daily for a period of 12 months. At Month 12, a post-treatment DBPCFC to peanut will be performed, with a starting dose of 1 mg peanut protein with escalation up to a highest dose of 2,000 mg peanut protein. This evaluation will help determine the primary efficacy endpoint of this pivotal study.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female children aged 4 through 11 years;
2. Physician-diagnosis of peanut allergy or children with a well documented medical history of IgE-mediated symptoms after ingestion of peanut and currently following a strict peanut-free diet, but without a physician diagnosis;
3. Peanut-specific IgE level (ImmunoCAP system) >0.7 kU/L;
4. Positive peanut skin prick test (SPT) with a largest wheal diameter:

   * ≥6 mm for children 4 through 5 years of age at Visit 1,
   * ≥8 mm for children 6 years and above at Visit 1;
5. Positive DBPCFC at ≤300 mg peanut protein.

Main Exclusion Criteria:

1. History of severe anaphylaxis to peanut with any of the following symptoms: hypotension, hypoxia, neurological compromise (collapse, loss of consciousness or incontinence);
2. Generalized dermatologic disease
3. Diagnosis of mast cell disorders, including mastocytosis or uricaria pigmentosa as well as hereditary or idiopathic angioedema;
4. Diagnosis of asthma that fulfills any of the following criteria:

   * Uncontrolled persistent asthma as defined by National Asthma Education and Prevention Program Asthma guidelines 2007 or by Global Initiative for Asthma guidelines 2015,
   * Asthma treated with either a high daily high dose of inhaled corticosteroid or with a combination therapy of a medium or high daily dose of inhaled corticosteroid with a long acting inhaled β2 agonist or with a combination therapy of a high daily dose of inhaled corticosteroid with a long acting inhaled β2 agonist. Asthmatic subjects treated with a medium daily dose of inhaled corticosteroids are eligible. Intermittent asthmatic subjects who require intermittent use of inhaled corticosteroids for rescue are also eligible,
   * Two or more systemic corticosteroid courses for asthma in the past year or 1 oral corticosteroid course for asthma within 3 months prior to Visit 1, or during screening period,
   * Prior intubation/mechanical ventilation for asthma within 1 year prior to Visit 1, or during screening;
5. Receiving β-blocking agents, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, calcium channel blockers or tricyclic antidepressant therapy;
6. Received anti-tumor necrosis factor drugs or anti-IgE drugs (such as omalizumab) or any biologic immunomodulatory therapy within 1 year prior to Visit 1, during screening period or during study participation;
7. Use of systemic long-acting corticosteroids within 12 weeks prior to Visit 1 and/or use of systemic short-acting corticosteroids within 4 weeks prior to Visit 1 or during screening;
8. Prior or concomitant history of any immunotherapy to any food;
9. Receiving or planning to receive any aeroallergen immunotherapy during their participation in the study. Aeroallergen immunotherapy must be discontinued at the time of Visit 1;
10. Any disorder in which epinephrine is contraindicated such as coronary artery disease, uncontrolled hypertension, or serious ventricular arrhythmias.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Fleischer, MD, Principal Investigator — Children's Hospital Colorado
Locations (31):
- United States (17):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, Rady Children's Hospital, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens' Hospital, Boston, Massachusetts
  - Jaffe Food Allergy Institute, New York, New York
  - The University of North Carolina - Chapell Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - ASTHMA, Inc., Seattle, Washington
- Australia (3):
  - Allergy Medical, Brisbane
  - Princess Margaret Hospital for Children, Perth
  - Children's Hospital Westmead, Sydney
- Canada (6):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Cheema Research Inc., Mississauga, Ontario
  - Ottawa Allergy Asthma Research Institute, Ottawa, Ontario
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - CHUM & CHU Sainte-Justine, Montreal, Quebec
  - Centre de Recherche Appliquée en Allergie de Québec (CRAAQ), Québec
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - St.-Marien-Hospital, Bonn
  - Universitätsklinikum Erlangen, Erlangen
- Ireland (2):
  - Clinical Investigations Unit, Cork
  - Our Lady's Children's Hospital, Dublin

REFERENCES:
- [Result] Fleischer DM, Greenhawt M, Sussman G, Begin P, Nowak-Wegrzyn A, Petroni D, Beyer K, Brown-Whitehorn T, Hebert J, Hourihane JO, Campbell DE, Leonard S, Chinthrajah RS, Pongracic JA, Jones SM, Lange L, Chong H, Green TD, Wood R, Cheema A, Prescott SL, Smith P, Yang W, Chan ES, Byrne A, Assa'ad A, Bird JA, Kim EH, Schneider L, Davis CM, Lanser BJ, Lambert R, Shreffler W. Effect of Epicutaneous Immunotherapy vs Placebo on Reaction to Peanut Protein Ingestion Among Children With Peanut Allergy: The PEPITES Randomized Clinical Trial. JAMA. 2019 Mar 12;321(10):946-955. doi: 10.1001/jama.2019.1113. PMID 30794314
- [Result] Greenhawt M, Kim EH, Campbell DE, Green TD, Lambert R, Fleischer DM. Improvements in eliciting dose across baseline sensitivities following 12 months of epicutaneous immunotherapy (EPIT) in peanut-allergic children aged 4 to 11 years. J Allergy Clin Immunol Pract. 2020 Oct;8(9):3219-3221. doi: 10.1016/j.jaip.2020.05.030. Epub 2020 Jun 2. No abstract available. PMID 32502548
- [Derived] Remington BC, Campbell DE, Green TD, Fleischer DM, Koppelman SJ. Post hoc analysis of epicutaneous immunotherapy for peanut allergy phase 3 results: Relevance for exposure through restaurant meals. Ann Allergy Asthma Immunol. 2021 Feb;126(2):208-209. doi: 10.1016/j.anai.2020.11.015. Epub 2020 Nov 28. No abstract available. PMID 33259921
- [Derived] Remington BC, Krone T, Kim EH, Bird JA, Green TD, Lack G, Fleischer DM, Koppelman SJ. Estimated risk reduction to packaged food reactions by epicutaneous immunotherapy (EPIT) for peanut allergy. Ann Allergy Asthma Immunol. 2019 Nov;123(5):488-493.e2. doi: 10.1016/j.anai.2019.08.007. Epub 2019 Aug 20. PMID 31442495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III study was conducted in participants aged 4 to 11 years old with peanut allergy at 31 active centers in Australia, Canada, Germany, Ireland and USA. Participants were randomized in a 2:1 ratio to receive DBV712 250 micrograms (μg) (Viaskin® Peanut 250 μg) or placebo.
Pre-assignment Details: A total of 500 participants signed an informed consent form and were enrolled in the study: 144 were screened failed and 356 were eligible and randomized in a 2:1 ratio to receive DBV712 250µg (n=238) or placebo (n=118).
  Maximum study duration for each participant was approximately 61 weeks (6-week screening period, 53-week treatment period and 2-week follow-up period).
Groups:
- DBV712 250 μg: Participants applied 1 new DBV712 250 μg patch for 24 hours (±4 hours) every day for 12 months. The application duration was progressively increased to a duration of 24 hours daily over a 15-day period (6 hours during the first week, 12 hours during the second week and 24 hours from the third week onwards).
- Placebo: Participants applied 1 new placebo patch for 24 hours (±4 hours) every day for 12 months. The application duration was progressively increased to a duration of 24 hours daily over a 15-day period (6 hours during the first week, 12 hours during the second week and 24 hours from the third week onwards).
- Screened: Total number of participant who signed an Informed Consent and were screened in the study to determine eligibility.
Period: Screening Period
Arm/Group | DBV712 250 μg | Placebo | Screened
Started | 0 | 0 | 500
Completed | 0 | 0 | 356
Not Completed | 0 | 0 | 144
Not completed — Inclusion/Exclusion Failure | 0 | 0 | 117
Not completed — Withdrawal by Subject | 0 | 0 | 23
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Other not specified | 0 | 0 | 3
Period: Treatment and Follow-up Periods
Arm/Group | DBV712 250 μg | Placebo | Screened
Started | 238 | 118 | 0
Completed | 213 | 107 | 0
Not Completed | 25 | 11 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0
Not completed — Non-compliance with the investigational product (IP) | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 13 | 6 | 0
Not completed — Other | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was comprised of all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | DBV712 250 μg | Placebo | Total
Number analyzed (Participants) | 238 | 118 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.4 (2.11) | 7.3 (2.30) | 7.3 (2.17)
Age, Customized [Count of Participants; unit: Participants]
  4 to 5 years | 55 | 32 | 87
  6 to 11 years | 183 | 86 | 269
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 49 | 138
  Male | 149 | 69 | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 194 | 96 | 290
  Black or African American | 1 | 2 | 3
  Asian | 19 | 8 | 27
  Other | 24 | 12 | 36
Screening Eliciting Dose (ED) Subgroup [Count of Participants; unit: Participants] — Screening ED Subgroup 1: participants with a screening ED of 1 mg, 3 mg or 10 mg peanut protein.
  Screening ED Subgroup 2: participants with a screening ED of 30 mg, 100 mg or 300 mg peanut protein.
  Participants
    Screening ED Subgroup 1 | 41 | 20 | 61
    Screening ED Subgroup 2 | 197 | 98 | 295

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentages of Treatment Responders at Month 12; Analyzed in the Overall Population
Description: The Double-Blind Placebo-Controlled Food Challenges (DBPCFCs) to determine Eliciting Dose (ED) were performed at screening and Month 12, with each challenge occurring over 2 days. The participant was gradually fed increasing amounts of standardized blinded oral formulas containing either peanut protein (during 1 of the 2 days of the challenge), or without any peanut protein (during the other day of the challenge). A participant was defined as a treatment responder if:
  * ED was ≥300 mg peanut protein at Month 12 DBPCFC (for screening ED subgroup 1), or
  * ED was ≥1,000 mg peanut protein at Month 12 DBPCFC (for screening ED subgroup 2).
  Participants with missing treatment response at Month 12 were imputed as non-responders. The percentage of treatment responders at Month 12 is presented. Analysis of the difference in response rates between treatment groups is presented in the subsequent statistical analysis table. Analysis was performed in the overall population.
Time Frame: At Month 12
Population: The Intent-to-Treat (ITT) population was comprised of all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DBV712 250 μg | Placebo
Number analyzed (Participants) | 238 | 118
percentage of participants | 35.3 [29.5 to 41.6] | 13.6 [8.5 to 20.9]
Statistical Analysis 1: Comparison: DBV712 250 μg vs Placebo; Analysis of the difference in response rates between DBV712 250 μg group and Placebo group and 2-sided Newcombe 95% confidence interval (CI). P-value was obtained from a 2-sided 5% test to evaluate the null hypothesis of no difference in response rates between treatment groups using the Wald method. Clinical relevance was evaluated based on the lower bound of the Newcombe 95% CI of the difference in response rates ≥15%; Test type: Other; p < 0.001, Wald; Difference in Response Rates (%) = 21.7, 95% CI 2-sided [12.4 to 29.8]

2. Secondary Outcome: Difference in Percentages of Treatment Responders at Month 12; Analyzed in Each Screening Eliciting Dose (ED) Subgroup
Description: The Double-Blind Placebo-Controlled Food Challenges (DBPCFCs) to determine Eliciting Dose (ED) were performed at screening and Month 12, with each challenge occurring over 2 days. The participant was gradually fed increasing amounts of blinded oral formulas containing either peanut protein (during 1 of the 2 days of the challenge), or without any peanut protein (during the other day of the challenge). A participant was defined as a treatment responder if:
  * ED was ≥300 mg peanut protein at Month 12 DBPCFC (for screening ED subgroup 1), or
  * ED was ≥1,000 mg peanut protein at Month 12 DBPCFC (for screening ED subgroup 2).
  Participants with missing treatment response at Month 12 were imputed as non-responders. The percentage of treatment responders at Month 12 is presented below. Analysis of the difference in response rates between treatment groups is presented in the subsequent statistical analysis table. Analysis was performed for each separate screening ED subgroup.
Time Frame: At Month 12
Population: The Intent-to-Treat (ITT) population was comprised of all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DBV712 250 μg | Placebo
Number analyzed (Participants) | 238 | 118
percentage of participants
  Screening ED subgroup 1: number analyzed (Participants) | 41 | 20
  Screening ED subgroup 1 | 39.0 [25.7 to 54.3] | 20.0 [8.1 to 41.6]
  Screening ED subgroup 2: number analyzed (Participants) | 197 | 98
  Screening ED subgroup 2 | 34.5 [28.2 to 41.4] | 12.2 [7.1 to 20.2]
Statistical Analysis 1: Comparison: DBV712 250 μg vs Placebo; Screening ED subgroup 1: Analysis of the difference in response rates between DBV712 250 μg group and Placebo group and 2-sided Newcombe 95% CI. P-value was obtained from a 2-sided 5% test to evaluate the null hypothesis of no difference in response rates between treatment groups using the Wald method. Clinical relevance was evaluated based on the lower bound of the Newcombe 95% CI of the difference in response rates >0; Test type: Other; p = 0.105, Wald; Difference in Response Rates (%) = 19.0, 95% CI 2-sided [-6.4 to 38.4]
Statistical Analysis 2: Comparison: DBV712 250 μg vs Placebo; Screening ED subgroup 2: Analysis of the difference in response rates between DBV712 250 μg group and Placebo group and 2-sided Newcombe 95% CI. P-value was obtained from a 2-sided 5% test to evaluate the null hypothesis of no difference in response rates between treatment groups using the Wald method. Clinical relevance was evaluated based on the lower bound of the Newcombe 95% CI of the difference in response rates >0; Test type: Other; p < 0.001, Wald; Difference in Response Rates (%) = 22.3, 95% CI 2-sided [12.1 to 30.8]

3. Secondary Outcome: Cumulative Reactive Dose (CRD) of Peanut Protein at Baseline and Month 12
Description: The CRD was calculated as the sum of all doses given (including any repeated and partial doses). The median CRD of peanut protein at baseline and Month 12 is presented. Analysis was performed using the modified baseline observation carried forward method to impute missing data at Month 12.
Time Frame: Baseline and Month 12
Population: The Intent-to-Treat (ITT) population was comprised of all participants who were randomized.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | DBV712 250 μg | Placebo
Number analyzed (Participants) | 238 | 118
mg
  Baseline | 144.0 [44.0 to 444.0] | 144.0 [44.0 to 444.0]
  Month 12 | 444.0 [144.0 to 1444.0] | 144.0 [44.0 to 444.0]
Statistical Analysis 1: Comparison: DBV712 250 μg vs Placebo; The treatment effect was estimated using the Hodges-Lehmann estimate of the difference in median CRDs at Month 12; Test type: Other; p < 0.001, Wilcoxon rank-sum test; Difference in Median CRD = 297.0, 95% CI 2-sided [130.0 to 317.0]

4. Other Pre Specified Outcome: Relative Change From Baseline in Peanut-specific Immunoglobulin E (IgE) Over Time
Description: Venous blood samples were drawn to assess peanut-specific IgE levels at baseline and Months 3, 6 and 12. The median relative changes from baseline in IgE levels for each timepoint are presented. Relative change from baseline=100×(value at the visit-value at baseline)/value at baseline.
Time Frame: Baseline and Months 3, 6 and 12
Population: The Intent-to-Treat (ITT) population was comprised of all participants who were randomized. Only those with non-missing data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Percent of change
Arm/Group | DBV712 250 μg | Placebo
Number analyzed (Participants) | 232 | 115
Percent of change
  Month 3 | 78.716 [26.557 to 174.588] | 16.964 [-12.591 to 48.802]
  Month 6: number analyzed (Participants) | 229 | 111
  Month 6 | 39.716 [-3.676 to 109.690] | 4.605 [-26.380 to 30.352]
  Month 12: number analyzed (Participants) | 224 | 108
  Month 12 | 2.858 [-24.739 to 61.058] | -6.919 [-31.468 to 25.291]

5. Other Pre Specified Outcome: Relative Changes From Baseline in Peanut-specific Immunoglobulin G4 Subtype (IgG4) Over Time
Description: Venous blood samples were drawn to assess peanut-specific IgG4 levels at baseline and Months 3, 6 and 12. The median relative changes from baseline in IgG4 levels for each timepoint are presented. Relative change from baseline=100×(value at the visit-value at baseline)/value at baseline.
Time Frame: Baseline and Months 3, 6 and 12
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percent of change
Arm/Group | DBV712 250 μg | Placebo
Number analyzed (Participants) | 231 | 115
Percent of change
  Month 3 | 127.778 [55.660 to 259.615] | 14.286 [0.000 to 45.833]
  Month 6: number analyzed (Participants) | 229 | 110
  Month 6 | 258.491 [107.843 to 549.351] | 11.492 [-9.677 to 42.105]
  Month 12: number analyzed (Participants) | 224 | 109
  Month 12 | 513.487 [196.458 to 1105.235] | 10.496 [-10.108 to 33.333]

ADVERSE EVENTS:
Time Frame: Screened arm: Adverse Events (AEs) collected from signing the informed consent up to the end of the screening period. DBV712 250µg and placebo arms: Treatment-Emergent Adverse Events (TEAEs) collected from Day 1, throughout the 53-week treatment period and additional 2-week follow-up period. Overall time frame of up to 55 weeks.
Description: Adverse Events were collected for the time the informed consent was signed up to the end of the study.
Groups:
- Screened: Participants enrolled in the study during the screening period prior randomization
Arm/Group | DBV712 250 μg | Placebo | Screened
All-Cause Mortality (participants affected / at risk) | 0/238 | 0/118 | 0/500
Serious Adverse Events (participants affected / at risk) | 10/238 | 6/118 | 9/500
Other Adverse Events (participants affected / at risk) | 222/238 | 96/118 | 83/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBV712 250 μg (N=238) | Placebo (N=118) | Screened (N=500)
Anaphylactic reaction (Immune system disorders) | 6 (7) | 3 (3) | 8 (8)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalitis influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBV712 250 μg (N=238) | Placebo (N=118) | Screened (N=500)
Upper respiratory tract infection (Infections and infestations) | 73 (134) | 30 (48) | 16 (16)
Viral upper respiratory tract infection (Infections and infestations) | 42 (82) | 20 (40) | 8 (8)
Gastroenteritis (Infections and infestations) | 20 (23) | 10 (11) | 2 (2)
Viral infection (Infections and infestations) | 19 (21) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 17 (20) | 3 (3) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 16 (23) | 5 (5) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 15 (17) | 3 (5) | 1 (1)
Influenza (Infections and infestations) | 7 (8) | 6 (6) | 2 (2)
Pyrexia (General disorders) | 48 (63) | 22 (34) | 5 (5)
Application site pruritus (General disorders) | 83 (154) | 14 (30) | 0 (0)
Application site erythema (General disorders) | 67 (118) | 20 (54) | 0 (0)
Application site swelling (General disorders) | 38 (86) | 2 (18) | 0 (0)
Application site eczema (General disorders) | 25 (29) | 6 (18) | 0 (0)
Application site reaction (General disorders) | 21 (29) | 2 (5) | 0 (0)
Application site urticaria (General disorders) | 16 (24) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 52 (97) | 15 (27) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 (78) | 16 (28) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 27 (50) | 9 (14) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 (34) | 10 (16) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 18 (26) | 9 (10) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (24) | 8 (12) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 27 (36) | 9 (31) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 21 (29) | 15 (25) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 18 (24) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 31 (42) | 10 (12) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 17 (19) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (18) | 3 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (16) | 7 (12) | 5 (5)
Food allergy (Immune system disorders) | 21 (29) | 9 (14) | 0 (0)
Hypersensitivity (Immune system disorders) | 22 (29) | 6 (8) | 4 (5)
Seasonal allergy (Immune system disorders) | 20 (30) | 5 (9) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 12 (12) | 4 (4) | 2 (2)
Allergy to animal (Immune system disorders) | 8 (11) | 8 (16) | 1 (1)
Headache (Nervous system disorders) | 39 (74) | 18 (41) | 5 (6)
Arthropod bite (Injury, poisoning and procedural complications) | 8 (9) | 6 (7) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT02636699/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT02636699/SAP_001.pdf